CLINICAL TRIAL: NCT05851378
Title: Hyperpolarized Carbon-13 Alpha-ketoglutarate Metabolic Imaging in IDH Mutant Glioma
Brief Title: Hyperpolarized Carbon-13 Alpha-ketoglutarate Imaging in IDH Mutant Glioma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Robert Bok, MD, PhD (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Robert Bok, MD, PhD, Participating Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 22925; NCI-2023-03744 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP)); 5P01CA118816-12 (NIH); 2P50CA097257 (NIH)
Record Dates: First submitted 2023-05-01; First posted 2023-05-09 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Adult Gliomas, Mixed
Keywords: Isocitrate Dehydrogenase Mutation
MeSH Terms: conditions — Glioma | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Hyperpolarized Carbon-13 Alpha-ketoglutarate (HP 13C-aKG) (Experimental): Cohort 1 will be comprised of 10 participants with Isocitrate dehydrogenase (IDH) mutant glioma who may or may not have received prior treatment for optimizing imaging protocol. Participants will be injected with 0.67ml/kg actual body weight of 100 millimolar (mM) of α-KG solution and have a single imaging scan.
- Cohort 2: Hyperpolarized Carbon-13 Alpha-ketoglutarate (HP 13C-aKG) (Experimental): Cohort 2 will be comprised 30 participants with recurrent IDH mutant glioma before receiving surgical resection. Participants will be injected with 0.67ml/kg actual body weight of 100 millimolar (mM) of α-KG solution and have a single imaging scan.

INTERVENTIONS:
Drug: Hyperpolarized Carbon 13 Alpha-ketoglutarate (HP C13-aKG) — Given intravenously at time of imaging
  Other Names: Hyperpolarized C13-aKG; HP C13-aKG
Procedure: Magnetic Resonance Image (MRI) — Magnetic resonance imaging is a medical imaging technique used in radiology to form pictures of the anatomy and the physiological processes of the body
  Other Names: MRI; MRI scan

SUMMARY:
This study will investigate the use of hyperpolarized (HP) carbon-13 (13C) alpha-ketoglutarate (aKG) (HP 13C-aKG) to characterize tumor burden in participants with isocitrate dehydrogenase (IDH) mutant glioma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To define the most appropriate imaging parameters for obtaining hyperpolarized 13C-aKG from participants with IDH mutant glioma.

II. To assess the safety and feasibility of hyperpolarized 13C-aKG magnetic resonance (MR) metabolic imaging as a new and unique tool for evaluating tumor burden in participants with IDH mutant glioma.

OUTLINE:

Participants will be assigned to one of 2 cohorts:

COHORT 1: Participants with IDH mutant glioma for sequence development.

COHORT 2: Participants with recurrent IDH mutant glioma before receiving surgical resection.

This imaging study will involve one MR scan with the administration of HP 13C-aKG and will receive a follow-up phone call within 1-7 days post-study to assess for late adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be > 18 years old who have evidence of evaluable disease (with contrast enhancing lesion or non-enhancing lesion > 1 cubic centimetre (cc))

* Cohort 1: Participants with IDH mutant glioma who may or may not have received prior treatment
* Cohort 2: Participants with recurrent IDH mutant glioma before receiving surgical resection,

All the subjects must have prior MR scans available for review to assess the location and size of residual/recurrent tumor and do not have contraindication for magnetic resonance (MR) examinations. To be included in the study all subjects must also meet the following criteria:

1. Participants must have a life expectancy > 8 weeks.
2. Participants must have a Karnofsky performance status of > 70.
3. Participants must have adequate renal function (creatinine < 1.5 mg/dL). This test must be performed within 60 days prior to the HP 13C Imaging scan.
4. Participants must not have any significant medical illnesses that in the investigator's opinion cannot be adequately controlled with appropriate therapy, would compromise the participant's ability to participate in this study or any disease that will obscure toxicity or dangerously impact response to the imaging agent.
5. Participants must not have New York Heart Association (NYHA) Grade II or greater congestive heart failure.
6. Participants must not have history of myocardial infarction or unstable angina within 12 months prior to study enrollment.
7. This study was designed to include women and minorities but was not designed to measure differences of intervention effects. Males and females will be recruited with no preference to gender. Minorities will actively be recruited to participate. No exclusion to this study will be based on race.
8. Participants must sign an informed consent indicating that they are aware of the investigational nature of this study. Participants must sign an authorization for the release of their protected health information.
9. Participants may not be known to be HIV-positive. HIV testing is not required for study participation.
10. Participants must not have a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless they are in complete remission and have been off all therapy for that disease for a minimum of 3 years.
11. Participants must not be pregnant or breast-feeding. Women of childbearing potential are required to obtain a negative pregnancy test within 14 days of Hyperpolarized Imaging scan. Effective contraception (men and women) must be used in subjects of childbearing potential.

Exclusion Criteria:

1. Participants are excluded from participating in this study if they are not able to comply with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-11 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Mean signal to noise ratio of HP 13C-aKG | Day of imaging (1 day)
  Signal-to-noise ratio (SNR) of HP 13C-aKG will be calculated voxel-by-voxel, and within each region of interest (ROI). The parameters considered will be the mean SNR, within these ROIs. Acquisition parameters will be optimized (such as spatial resolution) to have the highest metabolite SNR and metabolite contrast.
Mean signal to noise ratio of oncometabolite 2-hydroxyglutarate (2-HG) | Day of imaging (1 day)
  Signal-to-noise ratio (SNR) of HP 13C akG 2HG will be calculated voxel-by-voxel, and within each ROI. The parameters considered will be the mean SNR, the number of voxels with SNR 2HG within the normal brain > 3.0, the number of voxels with SNR 2HG within the lesion > 3.0. Acquisition parameters will be optimized (such as spatial resolution) to have the highest metabolite SNR and metabolite contrast. (2HG production only in the IDH mutant tumors).
Mean signal to noise ratio of of glutamate | Day of imaging (1 day)
  Signal-to-noise ratio (SNR) of 13C aKG glutamate will be calculated voxel-by-voxel, and within each region of interest. The parameters considered will be the number of voxels with SNR glutamate within the normal brain > 3.0, the number of voxels with SNR glutamate within the lesion > 3.0, Acquisition parameters will be optimized (such as spatial resolution) to have the highest metabolite SNR and metabolite contrast (reduced glutamate within the lesion compared to the normal brain).
Median signal to noise ratio of 2HG to aKG | Day of imaging (1 day)
  Metabolite ratios (2HG/aKG) will be calculated voxel-by-voxel, and within each ROI. Median, maximum, and sum of ratios will be reported. Acquisition parameters will be optimized (such as spatial resolution) to have the highest metabolite SNR and metabolite contrast (2HG production only in the IDH mutant tumors within the lesion compared to the normal brain).
Mean signal to noise ratio of 2HG to glutamate | Day of imaging (1 day)
  Metabolite ratios (2HG/glutamate) will be calculated voxel-by-voxel, and within each ROI. Median, maximum, and sum of ratios will be reported. Acquisition parameters will be optimized (such as spatial resolution) to have the highest metabolite SNR and metabolite contrast (2HG production only in the IDH mutant tumors and reduced glutamate within the lesion compared to the normal brain).
Proportion of participants who reported treatment-emergent adverse events | Day of imaging (1 day)
  Occurrence of clinically significant changes in safety variables, including injection site, as defined by the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be reported.
Comparison of HP 13C 2HG/aKG ratio with surgical results (Cohort 2) | Day of imaging (1 day)
  In Cohort 2, the ratio of 13C (2HG/aKG will be compared within normal appearing brain versus a brain with visible lesions using a two-sided paired t-test or Wilcoxon signed rank test
Comparison of HP 13C 2HG/glutamate ratio with surgical results (Cohort 2) | Day of imaging (1 day)
  In Cohort 2, the ratio of 13C 2HG/glutamate will be compared within a normal appearing brain versus a brain with visible lesions using a two-sided paired t-test or Wilcoxon signed rank test
Comparison of HP 13C glutamate/aKG ratio with surgical results (Cohort 2) | Day of imaging (1 day)
  In Cohort 2, the ratio of 13C glutamate/aKG will be compared within a normal appearing brain versus a brain with visible lesions using a two-sided paired t-test or Wilcoxon signed rank test

CONTACTS AND LOCATIONS:
Overall Officials: Susan Chang, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-10-18): https://cdn.clinicaltrials.gov/large-docs/78/NCT05851378/ICF_000.pdf